CLINICAL TRIAL: NCT06235385
Title: European Association of Cardiovascular Imaging Multiple and Mixed Valvular Disease Study
Acronym: EACVI-MMVD
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: European Association of Cardiovascular Imaging (Other)
Responsible Party: Sponsor
Other Study IDs: AP-HP : 231784
Record Dates: First submitted 2024-01-23; First posted 2024-01-31 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Heart Valve Diseases; Multiple Valve Disease, Unspecified; Aortic Valve Disease; Aortic Valve Stenosis; Aortic Valve Insufficiency; Mitral Valve Disease; Mitral Valve Stenosis; Mitral Valve Insufficiency and Aortic Valve Insufficiency; Mitral Valve Insufficiency; Aortic Valve Stenosis With Insufficiency; Mitral Valve Disease Mixed; Tricuspid Valve Insufficiency; Tricuspid Valve Disease; Tricuspid Stenosis
Keywords: Multiple Valvular Heart Disease; Mixed Valvular Heart Disease
MeSH Terms: conditions — Heart Valve Diseases; Aortic Valve Disease; Aortic Valve Stenosis; Aortic Valve Insufficiency; Mitral Valve Stenosis; Mitral Valve Insufficiency; Tricuspid Valve Insufficiency; Tricuspid Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Intervention not provided — This study is purely observational

SUMMARY:
This study aims to investigate the prevalence and characteristics of multiple and mixed valvular heart disease (MMVD), which includes combinations of stenotic or regurgitant lesions on cardiac valves. The research will be conducted as a multicenter observational study, involving several centers worldwide, and will have a one-year follow-up period (with a possible extension to 5 years). The primary aim is to determine the proportion of MMVD among patients evaluated for valvular heart disease. Secondary aims include the evaluation of the epidemiologic distribution of clinical, biological, and cardiovascular imaging characteristics at baseline, management strategies, and their impact on prognosis. The study will also evaluate clinical outcomes such as mortality, hospitalization for heart failure, and changes in echocardiographic parameters. This research aims to provide valuable insights into the diagnosis, management, and prognosis of MMVD, addressing an important knowledge gap in this area.

DETAILED DESCRIPTION:
Multiple and mixed valvular heart disease (MMVD), ie, the combination of stenotic or regurgitant lesions occurring on ≥2 cardiac valves (multiple valvular heart disease (VHD)) or the combination of stenotic and regurgitant lesions on the same valve (mixed VHD), are frequent in clinical routine. Nevertheless, their clinical, biological, cardiovascular imaging, and management is not well established.

This study will assess the proportion of MMVD including each combination of multiple and mixed VHD in a multicentre registry of all consecutive patients assessed on a cardiovascular imaging department for VHD. Furthermore, as secondary aims, baseline characteristics, decision-making and therapeutic strategy at baseline and their impact in terms of prognostic.

This is a prospective multicentre observational study involving 174 centres worldwide (35 countries) conducted as a cohort study with a 1-year follow-up (with possible extension to 5 years). Consecutive patients with a diagnosis of MMVD by echocardiography who meet the inclusion criteria will be included during the 6 months period of recruitment. In the context of a "real-life" cohort, baseline evaluation will be left to the discretion of the attending physician (and could encompass clinical evaluations, biomarkers, electrocardiograms, transthoracic and transoesophageal echocardiography, stress echocardiography, cardiac catheterization, invasive angiography, cardiac CT, and Cardiac MRI). Final diagnosis of the physician will be given, and physician will manage the patient in accordance with international guidelines (transcatheter valve intervention, surgery or no intervention). One year follow-up will be performed during a patient visit or by contact with the treating physician or the patient: vital status, hospitalizations for cardiac reasons (including heart failure), history of stroke and the performance of a new valvular intervention.

The primary endpoint will be the proportion of MMVD among all patients admitted for VHD evaluation in the imaging department. Secondary endpoints encompass; (i) epidemiologic distribution of clinical, biological, and cardiovascular imaging characteristics at baseline. (ii) proportion of MMVD treated by surgery, percutaneous or medical as well as the detail for management and how complication are managed (iii) prognostic evaluation at one year of follow-up in terms of clinical composite outcome (cardiovascular mortality, hospitalization for heart failure, myocardial infarction, pulmonary embolism and stroke), all-cause mortality, hospitalisation for heart failure, and change in echocardiographic parameters.

This is the first prospective multicentre study assessing the proportion of MMVD and their characteristics in term of diagnosis, management, and prognostic.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Patient referred to the cardiovascular imaging department.
3. Diagnosis of MMVD confirmed by transthoracic echocardiography, defined as:

   1. Multiple VHD: at least 2 moderates to severe VHD involving ≥ 2 different valves, using the current ESC guidelines.

      and/or
   2. Mixed VHD: at least moderate stenosis and at least moderate regurgitation of a single valve, using the current ESC guidelines.
4. Patient not refusing to have their data involved in the protocol after information.

Exclusion Criteria (patients fulfilling any of the following criteria are not eligible for inclusion in this study):

1. History of prior valve surgery or percutaneous valve intervention (concerning a valve other than those involved in the definition of MMVD).
2. Acute infective endocarditis at the time of evaluation for inclusion (confirmed according to modified Duke criteria) or history of endocarditis ≤ 6 months.
3. Complex congenital heart diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients referred to a Cardiovascular imaging Department with a diagnosis of at least one at least moderate VHD, and who meet the criteria for MMVD defined by multiple and/or mixed disease, will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of multiple and mixed valvular disease (MMVD) | Baseline
  Number of consecutive patients diagnosed with multiple and mixed valvular disease divided by the total number of consecutive patients assessed for valvular heart disease on a cardiovascular imaging department

SECONDARY OUTCOMES:
Major Adverse Cardiovascular Event (MACE) | Up to 5 years
  Clinical composite outcome defined as: cardiovascular mortality, hospitalization for heart failure (HF), myocardial infarction, pulmonary embolism and stroke.
All-cause mortality | Up to 5 years
  The adjudication of all-cause death was performed using the follow-up performed in clinical routine
Cardiovascular mortality | Up to 5 years
  The adjudication of cardiovascular mortality was performed using the follow-up performed in clinical routine
Hospitalization for heart failure | Up to 5 years
  Hospitalization for heart failure according to the European Society of Cardiology (ESC) guidelines

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hôpitaux de Paris, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No
Data cannot be shared for ethical/privacy reasons. The data cannot be shared publicly for the privacy of individuals that participated in the study and also because of regulatory constraints in the field of clinical research in France, it is unfortunately not possible to make the entire database available to all as an open source.

REFERENCES:
- [Derived] Unger A, Mandoli GE, Neglia D, Romero Dorta E, Kagiyama N, Borodzicz-Jazdzyk S, Velegraki E, Coisne A, Uygur B, Afana A, Florence J, Bohbot Y, Donal E, Clavel MA, Pibarot P, Unger P, Manka R, Nijveldt R, Gimelli A, Gerber B, Dweck M, Muraru D, Pontone G, Ajmone Marsan N, Timoteo AT, Toupin S, Pereira C, Cosyns B, Vicaut E, Delgado V, Petersen S, Pezel T. Rational and design of EACVI-MMVD study: an international registry on multimodality imaging for mixed and multiple valvular heart disease. Eur Heart J Imaging Methods Pract. 2026 Feb 2;4(1):qyaf156. doi: 10.1093/ehjimp/qyaf156. eCollection 2026 Jan. PMID 41635678